CLINICAL TRIAL: NCT04415411
Title: Effects of Nursing Care Provided to the Relatives of Palliative Care Patients on Caregivers' Spiritual Well-being and Hope: A Randomised Controlled Trial
Brief Title: Effects of Nursing Care Provided to Relatives of Palliative Care Patients on Caregivers' Spiritual Well-being and Hope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Asli Kurtgöz, PhD, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional; PYO. SBF.1904.19.006 (Other Grant/Funding Number: Ondokuz Mayıs University)
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Hope; Spirituality; Palliative Care
Keywords: family members; hope; nursing care; palliative care; spirituality; relatives

STUDY DESIGN:
Intervention Model Description: In this study, there are two groups as intervention group and control group. Investigator, administered not any application to control group. Nursing care which based on the Theory of Human Caring was given to intervention group for 4 weeks.
Masking Description: Due to the nature of the research, it was not possible to blind the participants to group assignment. Additionally, due to the study being conducted for a doctoral thesis, data collection (pre and posttest), interviews, interventions and evaluation of data carried out by the same researcher who was not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Routine nursing care
- Intervention group (Experimental): Nursing care based on the Theory of Human Caring
  Interventions: Other: Nursing care based on the Theory of Human Caring

INTERVENTIONS:
Other: Nursing care based on the Theory of Human Caring — Planned nursing care based on 10 caritas processes of Theory of Human Caring.
  Arms: Intervention group

SUMMARY:
The aim of this study is to determine the effects of nursing care provided based on the Watson's Theory of Human Caring to the relatives of palliative care patients on caregivers' spiritual well-being and hope. This research was conducted with 60 patient relatives (intervention group: 30, control group: 30) taking care of their patient in palliative care unit.

DETAILED DESCRIPTION:
Every year, millions of patients as well as millions of patients are primarily involved in the palliative care process. It is emphasized that from the very start of palliative care process until grievance stage, patient relatives require a myriad of physical, psychological, social and spiritual needs. It has been widely reported that among relatives of palliative care patients, there is a high incidence of mental distress, depression, anxiety, sleep disturbance, fear and despair. The maintain of hope and spiritual well-being are important in dealing with this difficult process. Accordingly, nursing care is important, which supports the hope and spiritual well-being of patients' relatives. Nursing care that supports hope and focuses on spiritual dimensions is important in Watson's Human Care Theory.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and above
* willingness and motivation to participate in research
* literacy
* being the primary caregiver
* lack of mental or verbal deficiency to respond the questions

Exclusion Criteria:

* aged 18 below
* unwilling to participate in research
* illiterate
* non-primary caregiver
* mental or communicative disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Hopeless level of patient relatives | 1. week
  Data were collected via Beck Hopelessness Scale. Maximum score to obtain from the scale varies in between 0-20. Higher scores obtained indicate that there is a high level of hopelessness in an individual.
Spiritual well-being level of patient relatives | 1. week
  Data were collected via Spiritual Well-Being Scale. Maximum score to obtain from the scale varies between 29-145. Higher score indicates stronger spiritual well-being.

SECONDARY OUTCOMES:
Hopeless level of patient relatives (Change in level of hopeless after 4 weeks) | 4 weeks
  Data were collected via Beck Hopelessness Scale. Maximum score to obtain from the scale varies in between 0-20. Higher scores obtained indicate that there is a high level of hopelessness in an individual.
Spiritual well-being level of patient relatives (Change in level of spiritual well-being after 4 weeks) | 4 weeks
  Data were collected via Spiritual Well-Being Scale. Maximum score to obtain from the scale varies between 29-145. Higher score indicates stronger spiritual well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Kurtgöz, PhD, Principal Investigator — Amasya University; Zeliha Koc, PhD, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans

REFERENCES:
- [Background] De Korte-Verhoef MC, Pasman HR, Schweitzer BP, Francke AL, Onwuteaka-Philipsen BD, Deliens L. Burden for family carers at the end of life; a mixed-method study of the perspectives of family carers and GPs. BMC Palliat Care. 2014 Mar 31;13(1):16. doi: 10.1186/1472-684X-13-16. PMID 24678941
- [Background] Gotze H, Brahler E, Gansera L, Polze N, Kohler N. Psychological distress and quality of life of palliative cancer patients and their caring relatives during home care. Support Care Cancer. 2014 Oct;22(10):2775-82. doi: 10.1007/s00520-014-2257-5. Epub 2014 May 9. PMID 24811216
- [Background] Ullrich A, Ascherfeld L, Marx G, Bokemeyer C, Bergelt C, Oechsle K. Quality of life, psychological burden, needs, and satisfaction during specialized inpatient palliative care in family caregivers of advanced cancer patients. BMC Palliat Care. 2017 May 10;16(1):31. doi: 10.1186/s12904-017-0206-z. PMID 28486962
- [Background] Oechsle K, Ullrich A, Marx G, Benze G, Heine J, Dickel LM, Zhang Y, Wowretzko F, Wendt KN, Nauck F, Bokemeyer C, Bergelt C. Psychological burden in family caregivers of patients with advanced cancer at initiation of specialist inpatient palliative care. BMC Palliat Care. 2019 Nov 18;18(1):102. doi: 10.1186/s12904-019-0469-7. PMID 31739802
- See also: WHO (2019). Palliative care — http://www.who.int/health-topics/palliative-care
- See also: Canadian Cancer Research Alliance (2017). Pan-canadian framework for palliative and end-of life care research — http://www.virtualhospice.ca/Assets/PEOLC_Report_EN(1)_20170605131142.pdf
- See also: Watson, J. (2010). Core concepts of Jean Watson's Theory of human caring/caring science. — http://www.watsoncaringscience.org/files/PDF/watsons-theory-of-human-caring-core-concepts-and-evolution-to-caritas-processes-handout.pdf